CLINICAL TRIAL: NCT01249989
Title: Make Better Choices (MBC) - Multiple Behavior Change in Diet and Activity
Brief Title: Make Better Choices
Acronym: MBC2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Bonnie Spring, Professor, Northwestern University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: R01HL075451 (NIH); R01HL075451 (NIH)
Record Dates: First submitted 2010-11-23; First posted 2010-11-30 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Health Behavior
Keywords: Physical Activity; Sedentary Lifestyle; Diet; Health Behavior
MeSH Terms: conditions — Health Behavior; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sequential MBC Condition (Experimental): Participants in the sequential condition will increase F/V consumption and decrease Sed behavior (weeks 1-6), then increase physical activity (weeks 7-12). Smartphones are equipped with customized real-time goal thermometers that provide objective feedback on target behaviors (FV, Sed, and PA). At the start of prescription, the FV and Sed goal thermometers are activated. During week 1-2, participants will close 1/3 of the gap between their baseline behaviors and target behaviors. During week 3-4 they will close 2/3 of the gap, and in weeks 5-6 they will achieve 100% of their goals. Participants will maintain these goals for the remainder of the 12-week intervention. At week 7, a real-time PA goal thermometer wirelessly linked to accelerometers will be activated. Similarly, in weeks 7-8 participants will be asked to close 1/3 of the gap between their baseline PA and target, in week 9-10 they will close 2/3 of the gap, and finally they will reach 100% of their PA goal in weeks 11-12.
  Interventions: Behavioral: Sequential MBC Condition
- Simultaneous MBC Condition (Experimental): Participants in the simultaneous condition will target FV+, Sed- and PA+ simultaneously. Participants will wear accelerometers and enter diet and sedentary activity 5 days/week on their Smartphone. All 3 goal thermometers will be activated from the outset of prescription (FV, Sed, PA). In week 1-2, participants will close 1/3 of the gap between their baseline FV, Sed, and PA behavior and their goals. In week 3-4 participants will close 2/3 of the gap, and 100% of their goals in weeks 5-6. Participants will maintain their target behaviors for FV, Sed and PA through week 12.
  Interventions: Behavioral: Simultaneous MBC Condition
- Stress Management Control (Active Comparator): Participants in the stress management control condition target stress, relaxation and sleep. This will serve as an attentional control condition. During the 12-week prescription period, participants will wear accelerometers, log hours slept, enter real-time information about their relaxation exercises and stress, and monitor 3 goal thermometers (sleep, relaxation, stress) to meet behavioral targets. Similarly, their goal is to close 1/3 of the gap between their baseline stress, sleep, and performance of relaxation exercises and the target criterion in weeks 1-2, close 2/3 of the gap in weeks 3-4, reach their targets in weeks 5-6, and then maintain these behavior changes through week 12.
  Interventions: Behavioral: Stress Management

INTERVENTIONS:
Behavioral: Sequential MBC Condition — Participants in the sequential condition will increase F/V consumption and decrease Sed behavior (weeks 1-6), then increase physical activity (weeks 7-12). Smartphones are equipped with customized real-time goal thermometers that provide objective feedback on target behaviors (FV, Sed, and PA). At the start of prescription, the FV and Sed goal thermometers are activated. During week 1-2, participants will close 1/3 of the gap between their baseline behaviors and target behaviors. During week 3-4 they will close 2/3 of the gap, and in weeks 5-6 they will achieve 100% of their goals. Participants will maintain these goals for the remainder of the 12-week intervention. At week 7, a real-time PA goal thermometer wirelessly linked to accelerometers will be activated. Similarly, in weeks 7-8 participants will be asked to close 1/3 of the gap between their baseline PA and target, in week 9-10 they will close 2/3 of the gap, and finally they will reach 100% of their PA goal in weeks 11-12.
  Arms: Sequential MBC Condition
Behavioral: Simultaneous MBC Condition — Simultaneous MBC condition will target FV+, Sed- and PA+ simultaneously. Participants in the simultaneous condition will wear their accelerometers and enter diet and sedentary activity 5 days/week. All 3 goal thermometers will be activated from the outset of prescription. The goal will be to close 1/3 of the gap between their FV, Sed, and PA statuses and the targets in weeks 1-2, close 2/3 of the gap in weeks 3-4, reach their targets in weeks 5-6, and then maintain target level behavior changes for FV, Sed and PA through week 12.
  Arms: Simultaneous MBC Condition
Behavioral: Stress Management — Participants in the stress management control condition target stress, relaxation and sleep. This will serve as an attentional control condition. During the 12-week prescription period, participants will wear accelerometers, log hours slept, enter real-time information about their relaxation exercises and stress, and monitor 3 goal thermometers (sleep, relaxation, stress) to meet behavioral targets. Similarly, their goal is to close 1/3 of the gap between their baseline stress, sleep, and performance of relaxation exercises and the target criterion in weeks 1-2, close 2/3 of the gap in weeks 3-4, reach their targets in weeks 5-6, and then maintain these behavior changes through week 12.
  Arms: Stress Management Control

SUMMARY:
The average adult has a poor quality diet and sedentary lifestyle, but the best way to produce sustained healthy change remains unknown. The MBC2 intervention uses handheld technology to help individuals monitor and transmit information about their eating and activity remotely to a behavior coach. The proposed trial tests whether MBC2 intervention improves diet and activity more than a stress management control condition, and whether changing multiple health behaviors is best achieved by changing them all at the same time, or one after another.

DETAILED DESCRIPTION:
Poor quality diet and physical inactivity are the most prevalent, preventable causes of death in the United States. In particular, high saturated fat diet (Fat), low fruit and vegetable intake (FV), low physical activity (PA), and high sedentary leisure screen time (Sed) co-occur and heighten the risks of cardiovascular disease and cancers. The first Make Better Choices (MBC1) experiment contrasted four strategies to promote healthful change across these four risk behaviors. Each intervention targeted two behaviors (one diet, one activity) simultaneously and either increased healthy or decreased unhealthy responding. The intervention targeting increased FV and decreased Sed was most efficacious, yielding unexpectedly sustained improvement in three out of the four risk behaviors (FV, Sed, Fat). The proposed MBC2 trial tests the efficacy of MBC intervention to promote sustained, healthful change in diet and activity at 6 and 12 months, as contrasted with a stress management control condition. MBC2 tests competing hypotheses about the optimal way to increase PA without undermining the maintenance of FV, Sed, and Fat by changing multiple behaviors either sequentially or simultaneously. Furthermore, MBC2 examines mediators and biomarkers of healthy lifestyle change. Community dwelling adults (N=250) with suboptimal diet and inactive lifestyle will be randomized to the following conditions: 1) Sequential MBC (increasing FV intake and decreasing Sed, followed by increasing PA), 2) Simultaneous MBC (increasing FV, decreasing Sed, and increasing PA), or 3) Control (stress management). Participants in all conditions will use Smartphones equipped with customized behavioral decision support tools to self-monitor health behaviors. These handheld devices will be programmed to automatically transmit these data to our study server to be reviewed by a personal behavior coach. Based on theories of self-regulation and habit strength, the Mastery hypothesis predicts superior health behavior change for participants randomized to the sequential condition. It is anticipated that these effects will be mediated by greater habit strength for healthy eating and physical activity. However, based on goal systems theory, the Synergy hypothesis predicts superior health behavior change among participants randomized to the simultaneous condition. It is anticipated that these effects will be mediated by the establishment of superordinate healthy lifestyle goals. The results of the MBC2 trial will assist researchers in understanding the optimal manner in which to facilitate multiple health behavior change in this population. Furthermore, these data will help to identify the mechanisms that underlie healthy change among prevalent risk behaviors. If successful, this trial will also result in an innovative, highly disseminable technology-supported minimal counseling intervention to address the American unhealthy diet and sedentary lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* Participants must expect to reside in the Chicagoland area for the next 9 months
* Must be willing to record diet, sedentary activities, and/or stress and sleep and wear an accelerometer for 12 weeks and intermittently thereafter for the next 9-months
* Must agree to make changes in eating and activity or in sleep and relaxation behaviors
* Participants must report all of the following on screening questionnaires:

  * Low fiber diet (< 9 FV servings/day)
  * High saturated fat intake (> 8% of daily calories from fat)
  * Less than 150 minutes per week of moderate intensity physical activity per week for the past 3 months (or less than 75 minutes of vigorous intensity activity per week)
  * An average of > 120 minutes/day spent on non-work, non-education related use of the following recreational sedentary pastimes: television, videos/movies, videogames, and computer use

Exclusion Criteria:

* Unstable medical conditions (e.g., uncontrolled hypertension, diabetes, recent myocardial infarction)
* Physician approval for those with existing and controlled medication conditions
* Those that require an assistive device for ambulation
* > 350 lbs
* Currently taking weight loss medications
* Psychiatric hospitalization in past 5 years
* Those at risk for adverse cardiovascular disease (CVD) events with moderate intensity activity (e.g., CVD symptoms while walking, those scheduled for cardiac stress test within 2 months)
* Those who cannot read English sufficiently to respond to self-report questionnaires
* Current or anticipated pregnancy
* Women who are lactating
* Current active eating disorders (anorexia, bulimia)
* Current substance abuse or dependence (other than nicotine)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2011-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in Fruit/Vegetable Serving Intake | 3, 6, and 9 months
  Change from baseline in standard fruit/vegetable serving intake measured at 3, 6, and 9 months.
Change in Saturated Fat (% of daily calories from fat) Intake | 3, 6, and 9-months
  Change from baseline in saturated fat intake (assessed by % of daily calories from fat) at 3, 6, 9-months.
Change in Sedentary Leisure Screen Time (minutes/week) | 3, 6, and 9-months
  Change from baseline in minutes per week of sedentary leisure screen time (e.g., TV watching, recreational computer use) at 3, 6, and 9-months.
Change in Physical Activity (minutes/week) | 3, 6, and 9-months
  Change from baseline in minutes per week of physical activity measured by accelerometer at 3, 6, and 9-months.
Change in Dietary Intake | 3 and 9-months
  Change from baseline in dietary consumption (e.g., fruits/vegetables) measured by clinician administered dietary recall (Block Food Frequency Questionnaire) at 3 and 9-months. This standardized measure will be used to validate the self-report data.
Healthy Diet and Activity Improvement | 3, 6, and 9 months
  Healthy diet and activity improvement standardized to a common z score metric and aggregated across changes in fruit and vegetable intake, saturated fat intake, sedentary leisure screen time, and physical activity

SECONDARY OUTCOMES:
Change in Blood Pressure (mmHg) | 3 and 9-months
  Change from baseline in blood pressure measured in mmHg according to the CARDIA protocol.
Change in Lipids | 3 and 9-months
  Change from baseline in lipids (total cholesterol, triglycerides, HDL-C, calculated LDL-C) assayed following antecubital venipuncture
Change in Insulin (mg/dL) | 3 and 9-months
  Change from baseline in insulin measured in mg/dL via immunoassay following antecubital venipuncture at 3 and 9-months.
Change in Weight (kg) | 3 and 9-months
  Change from baseline in body weight in kg measured using calibrated beam balance scale at 3 and 9-months.
Change in Waist circumference (cm) | 3 and 9-months
  Change from baseline in waist circumference measured in cm (repeated twice, then averaged) at 3 and 9-months.
Change in Quality of Life | 3 and 9-months
  Change from baseline in quality of life measured by the SF-36 self-report questionnaire at 3 and 9-months.

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Spring, PhD, ABPP, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University-Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pellegrini CA, Steglitz J, Johnston W, Warnick J, Adams T, McFadden HG, Siddique J, Hedeker D, Spring B. Design and protocol of a randomized multiple behavior change trial: Make Better Choices 2 (MBC2). Contemp Clin Trials. 2015 Mar;41:85-92. doi: 10.1016/j.cct.2015.01.009. Epub 2015 Jan 24. PMID 25625810
- [Derived] Hibler E, Huang L, Andrade J, Spring B. Impact of a diet and activity health promotion intervention on regional patterns of DNA methylation. Clin Epigenetics. 2019 Sep 11;11(1):133. doi: 10.1186/s13148-019-0707-0. PMID 31506096
- [Derived] Spring B, Pellegrini C, McFadden HG, Pfammatter AF, Stump TK, Siddique J, King AC, Hedeker D. Multicomponent mHealth Intervention for Large, Sustained Change in Multiple Diet and Activity Risk Behaviors: The Make Better Choices 2 Randomized Controlled Trial. J Med Internet Res. 2018 Jun 19;20(6):e10528. doi: 10.2196/10528. PMID 29921561